CLINICAL TRIAL: NCT02485158
Title: A Preliminary Investigation of Individual Differences in Subjective Responses to D-amphetamine, Alcohol, and Delta-9-tetrahydrocannabinol
Brief Title: Individual Differences in the Response to Drugs
Acronym: TDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB13-0534
Record Dates: First submitted 2015-06-24; First posted 2015-06-30 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Subjective Effects; Alcohol; Amphetamine; THC; Personality
MeSH Terms: interventions — Dronabinol; Adenosine Monophosphate; Dextroamphetamine; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMP, ALC, THC or Placebo 1 (Experimental): All healthy adult volunteers attended 6 sessions in which they received 20mg AMP, 0.8g/kg ALC, and 7.5mg THC, alternating with three placebo sessions.
  Interventions: Drug: THC; Drug: AMP; Drug: ALC; Drug: Placebo capsules; Drug: Placebo beverage
- AMP, ALC, THC or Placebo 2 (Experimental): All healthy adult volunteers attended 6 sessions in which they received 20mg AMP, 0.8g/kg ALC, and 7.5mg THC, alternating with three placebo sessions.
  Interventions: Drug: THC; Drug: AMP; Drug: ALC; Drug: Placebo capsules; Drug: Placebo beverage

INTERVENTIONS:
Drug: THC — This is a within-subjects, double-blind, placebo controlled design. We administered oral THC to healthy volunteers to measure their subjective response, which we later compared to their responses to two other drugs.
  Other Names: delta-9-tetrahydrocannabinol
Drug: AMP — This is a within-subjects, double-blind, placebo controlled design. We administered AMP to healthy volunteers to measure their subjective response, which we later compared to their responses to two other drugs.
  Other Names: d-Amphetamine
Drug: ALC — This is a within-subjects, double-blind, placebo controlled design. We administered alcohol to healthy volunteers to measure their subjective response, which we later compared to their responses to two other drugs.
  Other Names: Alcohol
Drug: Placebo capsules — This is a within-subjects, double-blind, placebo controlled design. We administered size 00 gelatin capsules containing dextrose to healthy volunteers as a control for when they received either amphetamine or THC.
  Other Names: Sugar Pills
Drug: Placebo beverage — This is a within-subjects, double-blind, placebo controlled design. We administered a drink containing cranberry juice plus 1% alcohol added as a taste mask.

SUMMARY:
The purpose of this study is to examine whether individual differences in acute responses to drugs co-vary across three drugs from different drug classes: alcohol, amphetamine and delta-9-tetrahydrocannabinol (THC). The investigators hypothesize that individuals who experience greater rewarding effects from one drug will also experience more rewarding effects from the other drugs.

DETAILED DESCRIPTION:
Here, the investigators aim to investigate whether individuals exhibit similar responses to three different drugs from different classes. This study used a within-subjects design (total N = 24). All subjects received alcohol, amphetamine and delta-9-tetrahydrocannabinol (THC) in a double-blind, double-dummy fashion. Subjects completed six sessions wherein they received either alcohol, amphetamine, or THC, or corresponding placebos, on separate days. Subjects completed questionnaires about mood, general drug effects, and specific drug effects.

ELIGIBILITY:
Inclusion Criteria:

* English fluency
* High school education
* BMI between 19 and 26
* Individuals who report drinking at least 4 alcoholic drinks on one occasion in the past month

Exclusion Criteria:

* individuals with a medical condition contraindicating study participation, as determined by our physician
* individuals regularly using any contraindicated medications
* individuals with current dependence on any drug or past dependence on alcohol, marijuana or stimulants
* individuals with a past year DSM-IV Axis I mood, anxiety, eating, or psychotic disorder
* women who are pregnant, nursing, or planning to become pregnant in the next 3 months
* individuals who drink more than 10 alcoholic drinks per week
* individuals who currently use i) any illicit drug weekly or more frequently, ii) stimulant prescription drugs, iii) more than 10 cigarettes per week, and iv) more than 3 cups of coffee per day

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet de Wit, PhD, Principal Investigator — University of Chicago

REFERENCES:
- [Derived] Wardle MC, Marcus BA, de Wit H. A Preliminary Investigation of Individual Differences in Subjective Responses to D-Amphetamine, Alcohol, and Delta-9-Tetrahydrocannabinol Using a Within-Subjects Randomized Trial. PLoS One. 2015 Oct 29;10(10):e0140501. doi: 10.1371/journal.pone.0140501. eCollection 2015. PMID 26513587

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy social drinkers were recruited from the Chicago area through flyers and online advertisements, from June 2013 through February 2014.
Groups:
- Healthy Adult Volunteers: 24 healthy adult volunteers completed a 6 session within-subject, double-blind, placebo-controlled trial. At three of these sessions, they received one of three recreational drugs, d-amphetamine, THC and alochol (only one drug was administered per drug session). The other three sessions were matched placebo sessions. At each session, they received a capsule and a drink. At the amphetamine drug session, they received a capsule containing d-amphetamine and a placebo beverage. At the THC drug session, they received a capsule containing THC and a placebo beverage. At the alcohol drug session they received a placebo capsule and a beverage containing alcohol. At the three matched placebo sessions, both the capsule and the beverage were placebo.
Period: Overall Study
Arm/Group | Healthy Adult Volunteers
Started | 28
Completed | 24
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — expected drug side effect | 1

BASELINE CHARACTERISTICS:
Groups:
- Healthy Adult Volunteers: All healthy adult volunteers completed a 6 session within-subject, double-blind, placebo-controlled trial. At three of these sessions, they received one of three recreational drugs, d-amphetamine, THC and alochol (only one drug was administered per drug session). The other three sessions were matched placebo sessions. At each session, they received a capsule and a drink. At the amphetamine drug session, they received a capsule containing d-amphetamine and a placebo beverage. At the THC drug session, they received a capsule containing THC and a placebo beverage. At the alcohol drug session they received a placebo capsule and a beverage containing alcohol. At the three matched placebo sessions, both the capsule and the beverage were placebo.
Arm/Group | Healthy Adult Volunteers
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.6 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in General Drug Effects (Drug Effects Questionnaire) at 30 Minutes After Capsule Administration
Description: Drug effects will be measured using the Drug Effects Questionnaire (Fischman & Foltin, 1991). The DEQ included 5 subscales; feeling, liking, and disliking the drug effect, feeling high, and wanting more of the drug. Each subscale ranged from 1(Not at all) to 100(Very much). The change in DFQ was assessed by the difference in measurements between baseline and 30 minutes after capsule administration and before drink administration. Baseline was measure 15 minutes prior to capsule administration.
Time Frame: Measured 15 minutes prior to capsule administration and 30 minutes after capsule administration and before drink administration
Population: Participants who completed all sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- AMP Arm: All healthy adult volunteers completed a 6 session; The three recreational drugs, d-amphetamine, THC and alochol (only one drug was administered per drug session). The other three sessions were matched placebo sessions. AMP arm represents a amphetamine drug session in which participants received a capsule containing d-amphetamine.
- ALC Arm: All healthy adult volunteers completed a 6 session; The three recreational drugs, d-amphetamine, THC and alochol (only one drug was administered per drug session). The other three sessions were matched placebo sessions. ALC arm represents a session in which participants received alcohol beverage.
- THC Arm: All healthy adult volunteers completed a 6 session; The three recreational drugs, d-amphetamine, THC and alochol (only one drug was administered per drug session). The other three sessions were matched placebo sessions. At the THC drug session, they received a capsule containing THC.
- AMP Placebo Arm: All healthy adult volunteers completed a 6 session; The three recreational drugs, d-amphetamine, THC and alochol (only one drug was administered per drug session). The other three sessions were matched placebo sessions. AMP placebo arm represents a session in which participants received a placebo drug.
- ALC Placebo Arm: All healthy adult volunteers completed a 6 session; The three recreational drugs, d-amphetamine, THC and alochol (only one drug was administered per drug session). The other three sessions were matched placebo sessions. ALC placebo arm represents a session in which participants received a placebo beverage.
- THC Placebo Arm: All healthy adult volunteers completed a 6 session; The three recreational drugs, d-amphetamine, THC and alochol (only one drug was administered per drug session). The other three sessions were matched placebo sessions. THC placebo arm represents a session in which participants received a placebo drug.
Arm/Group | AMP Arm | ALC Arm | THC Arm | AMP Placebo Arm | ALC Placebo Arm | THC Placebo Arm
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  DEQ Feel | 4.79 (7.22) | 12.83 (18.78) | 11.08 (21.09) | 12.17 (19.90) | 9.38 (11.12) | 4.5 (13.16)
  DEQ Like | 16.08 (27.47) | 18.67 (28.81) | 11.75 (21.84) | 9.0 (18.42) | 10.04 (17.90) | 9.67 (24.14)
  DEQ Dislike | 4.21 (9.43) | 11.71 (20.35) | 12.38 (23.77) | 10.71 (18.75) | 11.0 (20.60) | 0.83 (2.24)
  DEQ High | 3.29 (6.06) | 8.83 (16.31) | 10.58 (21.85) | 6.96 (18.44) | 5.5 (10.43) | 3.67 (9.40)
  DEQ More | 14.21 (25.26) | 13.5 (25.24) | 6.54 (13.71) | 5.63 (12.59) | 3.71 (7.66) | 11.0 (25.32)

2. Primary Outcome: Change in General Drug Effects (Drug Effects Questionnaire) at 30 Minutes After Drink Administration
Description: Drug effects will be measured using the Drug Effects Questionnaire (Fischman & Foltin, 1991). The DEQ included 5 subscales; feeling, liking, and disliking the drug effect, feeling high, and wanting more of the drug. Each subscale ranged from 1(Not at all) to 100(Very much). The change in DFQ was assessed by the difference in measurements between baseline and 30 minutes after drink administration. Baseline was measure 15 minutes prior to capsule administration.
Time Frame: Measured 15 minutes prior to capsule administration and 30 minutes after drink administration.
Population: Participants who completed all sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMP Arm | ALC Arm | THC Arm | AMP Placebo Arm | ALC Placebo Arm | THC Placebo Arm
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  DEQ Feel | 43.42 (29.53) | 76.83 (20.01) | 38.25 (33.45) | 21.58 (19.52) | 17.83 (22.56) | 18.63 (20.69)
  DEQ Like | 53.88 (34.49) | 45.08 (28.43) | 28.75 (30.05) | 16.63 (22.89) | 14.38 (20.78) | 25.29 (28.76)
  DEQ Dislike | 15.71 (22.76) | 43.96 (28.96) | 25.63 (35.03) | 17.71 (23.32) | 16.68 (26.83) | 15.79 (20.66)
  DEQ High | 30.5 (27.78) | 50.38 (32.15) | 31.75 (35.00) | 12.54 (18.09) | 11.5 (21.80) | 12.96 (20.22)
  DEQ More | 42.17 (35.27) | 24.75 (32.67) | 17.46 (25.18) | 10.96 (19.14) | 10.0 (18.32) | 18.96 (28.97)

3. Primary Outcome: Change in General Drug Effects (Drug Effects Questionnaire) at 90 Minutes After Drink Administration
Description: Drug effects will be measured using the Drug Effects Questionnaire (Fischman & Foltin, 1991). The DEQ included 5 subscales; feeling, liking, and disliking the drug effect, feeling high, and wanting more of the drug. Each subscale ranged from 1(Not at all) to 100(Very much). The change in DFQ was assessed by the difference in measurements between baseline and 90 minutes after drink administration. Baseline was measure 15 minutes prior to capsule administration.
Time Frame: Measured 15 minutes prior to capsule administration and 90 minutes after drink administration.
Population: Participants who completed all sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMP Arm | ALC Arm | THC Arm | AMP Placebo Arm | ALC Placebo Arm | THC Placebo Arm
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  DEQ Feel | 34.92 (24.75) | 61.21 (24.02) | 31.54 (31.41) | 16.46 (18.97) | 12.75 (18.74) | 13.17 (19.05)
  DEQ Like | 55.67 (31.45) | 29.92 (28.57) | 20.08 (26.32) | 10.42 (18.22) | 11.38 (19.35) | 13.25 (22.87)
  DEQ Dislike | 16.54 (21.60) | 50.46 (26.47) | 23.25 (29.72) | 17.54 (26.16) | 15.33 (24.85) | 15.96 (24.91)
  DEQ High | 27.92 (24.57) | 41.83 (30.74) | 29.21 (32.78) | 6.83 (12.47) | 7.25 (13.50) | 7.58 (12.65)
  DEQ More | 50.21 (36.06) | 25.88 (35.11) | 16.54 (23.69) | 6.54 (15.33) | 7.71 (16.59) | 12.88 (21.88)

4. Primary Outcome: Change in General Drug Effects (Drug Effects Questionnaire) at 120 Minutes After Drink Administraion
Description: Drug effects will be measured using the Drug Effects Questionnaire (Fischman & Foltin, 1991). The DEQ included 5 subscales; feeling, liking, and disliking the drug effect, feeling high, and wanting more of the drug. Each subscale ranged from 1(Not at all) to 100(Very much). The change in DFQ was assessed by the difference in measurements between baseline and 120 minutes after drink administration. Baseline was measure 15 minutes prior to capsule administration.
Time Frame: Measured 15 minutes prior to capsule administration and 120 minutes after drink administration.
Population: Participants who completed all sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMP Arm | ALC Arm | THC Arm | AMP Placebo Arm | ALC Placebo Arm | THC Placebo Arm
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  DEQ Feel | 27.08 (22.38) | 43.92 (24.18) | 24.08 (29.28) | 11.92 (14.26) | 7.96 (14.08) | 7.88 (14.65)
  DEQ Like | 43.75 (36.08) | 23.79 (25.61) | 18 (27.26) | 7.04 (13.90) | 4.83 (11.49) | 8.67 (16.86)
  DEQ Dislike | 11.92 (19.56) | 44.92 (31.37) | 19.63 (27.21) | 13.38 (22.39) | 11.08 (23.89) | 8.88 (18.69)
  DEQ High | 18.88 (21.43) | 29.38 (25.77) | 21.96 (30.06) | 5.04 (8.12) | 5.08 (11.20) | 4.83 (10.45)
  DEQ More | 45.38 (34.86) | 17.5 (27.95) | 9.92 (18.06) | 3.13 (5.53) | 6.54 (15.59) | 9.88 (19.63)

5. Primary Outcome: Change in General Drug Effects (Drug Effects Questionnaire) at 150 Minutes After Drink Administration
Description: Drug effects will be measured using the Drug Effects Questionnaire (Fischman & Foltin, 1991). The DEQ included 5 subscales; feeling, liking, and disliking the drug effect, feeling high, and wanting more of the drug. Each subscale ranged from 1(Not at all) to 100(Very much). The change in DFQ was assessed by the difference in measurements between baseline and 150 minutes after drink administration. Baseline was measure 15 minutes prior to capsule administration.
Time Frame: Measured 15 minutes prior to capsule administration and 150 minutes after drink administration.
Population: Participants who completed all sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMP Arm | ALC Arm | THC Arm | AMP Placebo Arm | ALC Placebo Arm | THC Placebo Arm
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  DEQ Feel | 19.79 (17.72) | 30.83 (22.52) | 18.63 (25.28) | 5.83 (10.72) | 4.63 (10.48) | 4.63 (7.80)
  DEQ Like | 39.5 (34.58) | 21.33 (24.74) | 11.71 (19.22) | 6.74 (14.88) | 2.42 (6.76) | 4.96 (14.48)
  DEQ Dislike | 11.25 (20.64) | 40.75 (32.31) | 17.79 (26.78) | 8.09 (21.80) | 4.29 (13.84) | 6.42 (15.69)
  DEQ High | 16.33 (18.68) | 20.46 (23.70) | 14.75 (20.27) | 2.87 (4.48) | 2.13 (4.83) | 1.96 (4.56)
  DEQ More | 44.08 (34.63) | 12.58 (24.39) | 9.38 (18.95) | 2.87 (10.55) | 5.04 (12.75) | 6.21 (15.19)

6. Primary Outcome: Change in General Drug Effects (Drug Effects Questionnaire) at 180 Minutes After Drink Administration
Description: Drug effects will be measured using the Drug Effects Questionnaire (Fischman & Foltin, 1991). The DEQ included 5 subscales; feeling, liking, and disliking the drug effect, feeling high, and wanting more of the drug. Each subscale ranged from 1(Not at all) to 100(Very much). The change in DFQ was assessed by the difference in measurements between baseline and 180 minutes after drink administration. Baseline was measure 15 minutes prior to capsule administration.
Time Frame: Measured 15 minutes prior to capsule administration and 180 minutes after drink administration.
Population: Participants who completed all sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMP Arm | ALC Arm | THC Arm | AMP Placebo Arm | ALC Placebo Arm | THC Placebo Arm
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  DEQ Feel | 16.13 (17.06) | 22.21 (19.71) | 15.67 (24.63) | 3.5 (8.548) | 2.08 (5.01) | 2.54 (4.59)
  DEQ Like | 31.08 (34.86) | 9.04 (14.29) | 7.33 (15.82) | 2.54 (11.23) | 1.75 (7.56) | 4.0 (12.47)
  DEQ Dislike | 11.54 (25.17) | 29.5 (34.28) | 16.13 (28.42) | 4.25 (17.24) | 4.29 (16.80) | 4.63 (13.65)
  DEQ High | 11.67 (15.29) | 14.13 (19.36) | 11.79 (18.36) | 1.63 (4.92) | 1.25 (3.30) | 1.04 (3.30)
  DEQ More | 38.38 (34.54) | 7.0 (19.77) | 10.04 (18.61) | 2.46 (10.99) | 4.04 (12.22) | 5.04 (12.89)

7. Primary Outcome: Change in General Drug Effects (Drug Effects Questionnaire) at 210 Minutes After Drink Administration
Description: Drug effects will be measured using the Drug Effects Questionnaire (Fischman & Foltin, 1991). The DEQ included 5 subscales; feeling, liking, and disliking the drug effect, feeling high, and wanting more of the drug. Each subscale ranged from 1(Not at all) to 100(Very much). The change in DFQ was assessed by the difference in measurements between baseline and 210 minutes after drink administration. Baseline was measure 15 minutes prior to capsule administration.
Time Frame: Measured 15 minutes prior to capsule administration and 210 minutes after drink administration.
Population: Participants who completed all sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMP Arm | ALC Arm | THC Arm | AMP Placebo Arm | ALC Placebo Arm | THC Placebo Arm
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  DEQ Feel | 11.08 (16.71) | 12.88 (15.88) | 5.79 (10.91) | 2.17 (5.74) | 0.96 (2.74) | 1.08 (2.75)
  DEQ Like | 18.38 (31.38) | 7.33 (14.62) | 4.88 (10.41) | 1.96 (7.04) | 0.25 (0.74) | 4.38 (13.73)
  DEQ Dislike | 8.54 (24.16) | 22.71 (30.79) | 6.83 (15.46) | 7.46 (23.16) | 1.29 (3.82) | 4.54 (15.14)
  DEQ High | 6.25 (9.88) | 9.21 (15.84) | 4.96 (11.02) | 0.33 (1.05) | 0.83 (1.76) | 0.42 (1.32)
  DEQ More | 32.5 (31.84) | 4.54 (17.72) | 8.79 (17.04) | 2.25 (8.19) | 3.83 (12.09) | 6.17 (14.65)

8. Primary Outcome: Change in Specific Drug Effects (Addiction Research Center Inventory) at 30 Minutes After Capsule Administration
Description: Specific drug effects will be measured using the Addiction Research Center Inventory (Martin et al. 1971). The ARCI measures effects specific to drug classes, including the effects of AMP-like drugs (A scale, 0 to 11), morphine and benzedrine like drugs (MBG scale, 0 to 14), lysergic acid-like drugs (LSD scale, 0 to 14), benzedrine-like drugs (BG scale, 0 to 13), pentobarbital-chlorpromazine and ALC-like drugs (PCAG scale, 0 to 15), and cannabis-like drugs (M scale, 0 to 12). We used this questionnaire as a manipulation check to ensure that the drugs produced their typical drug-specific effects in this study. For example, zero value of A sacle would be minimum report of amphetamine-like drug effects, and 11 would be maximum report of amphetamine-like effects. The change in ARCI was assessed by the difference in measurements between baseline and 30 minutes after capsule administration and before drink administration. Baseline was measure 15 minutes prior to capsule administration.
Time Frame: as for outcome 1
Population: Participants who completed all sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMP Arm | ALC Arm | THC Arm | AMP Placebo Arm | ALC Placebo Arm | THC Placebo Arm
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  ARC A | -0.17 (0.92) | 0.25 (1.33) | -0.04 (1.16) | -0.25 (0.61) | -0.17 (1.2) | 0.54 (0.88)
  ARC MBG | -0.58 (1.44) | -0.29 (1.27) | -0.71 (1.88) | -0.58 (0.65) | -0.67 (1.46) | 0.33 (1.37)
  ARC LSD | 0.13 (0.85) | 0.33 (0.82) | 0.38 (1.69) | 0.13 (0.99) | 0.08 (0.97) | -0.17 (0.64)
  ARC BG | -0.46 (1.02) | -0.75 (1.67) | -0.79 (2.0) | -1.17 (1.52) | -0.92 (1.21) | 0.25 (1.03)
  ARC PCAG | 0.58 (1.21) | 1.29 (2.39) | 2.92 (2.73) | 1.96 (2.44) | 0.92 (1.61) | 0.42 (1.02)
  ARC M | 0.08 (1.06) | 0.83 (1.81) | 0.42 (1.32) | 0.5 (1.25) | 0.33 (1.05) | 0.42 (1.18)

9. Primary Outcome: Change in Specific Drug Effects (Addiction Research Center Inventory) at 30 Minutes After Drink Administration
Description: Specific drug effects will be measured using the Addiction Research Center Inventory (Martin et al. 1971). The ARCI measures effects specific to drug classes, including the effects of AMP-like drugs (A scale, 0 to 11), morphine and benzedrine like drugs (MBG scale, 0 to 14), lysergic acid-like drugs (LSD scale, 0 to 14), benzedrine-like drugs (BG scale, 0 to 13), pentobarbital-chlorpromazine and ALC-like drugs (PCAG scale, 0 to 15), and cannabis-like drugs (M scale, 0 to 12). We used this questionnaire as a manipulation check to ensure that the drugs produced their typical drug-specific effects in this study. For example, zero value of A sacle would be minimum report of amphetamine-like drug effects, and 11 would be maximum report of amphetamine-like effects. The change in ARCI was assessed by the difference in measurements between baseline and 30 minutes after drink administration. Baseline was measure 15 minutes prior to capsule administration.
Time Frame: Measured 15 minutes prior to capsule administration and 30 minutes after drink administration
Population: Participants who completed all sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMP Arm | ALC Arm | THC Arm | AMP Placebo Arm | ALC Placebo Arm | THC Placebo Arm
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  ARC A | 2.88 (2.80) | 1.92 (2.64) | 0.17 (0.96) | 0 (0.93) | -0.33 (1.61) | 0.71 (1.40)
  ARC MBG | 3.71 (4.59) | 1.38 (4.79) | -0.54 (3.04) | 0 (1.77) | -1.17 (2.75) | 0.88 (3.26)
  ARC LSD | 1.13 (2.03) | 2.63 (2.32) | 1.54 (2.47) | 0.33 (1.09) | 0.29 (1.12) | 0.13 (1.23)
  ARC BG | 1.63 (2.28) | -0.88 (3.00) | -1.38 (1.64) | -0.83 (1.31) | -0.96 (1.99) | 0.04 (1.46)
  ARC PCAG | -1 (1.89) | 3.71 (4.29) | 2.96 (3.33) | 2.25 (3.55) | 1.54 (3.24) | 1.13 (2.35)
  ARC M | 3.21 (2.73) | 3.42 (2.22) | 2.04 (2.56) | 0.42 (0.93) | 0.29 (1.16) | 0.96 (1.78)

10. Primary Outcome: Change in Specific Drug Effects (Addiction Research Center Inventory) at 90 Minutes After Drink Administration
Description: Specific drug effects will be measured using the Addiction Research Center Inventory (Martin et al. 1971). The ARCI measures effects specific to drug classes, including the effects of AMP-like drugs (A scale, 0 to 11), morphine and benzedrine like drugs (MBG scale, 0 to 14), lysergic acid-like drugs (LSD scale, 0 to 14), benzedrine-like drugs (BG scale, 0 to 13), pentobarbital-chlorpromazine and ALC-like drugs (PCAG scale, 0 to 15), and cannabis-like drugs (M scale, 0 to 12). We used this questionnaire as a manipulation check to ensure that the drugs produced their typical drug-specific effects in this study. For example, zero value of A sacle would be minimum report of amphetamine-like drug effects, and 11 would be maximum report of amphetamine-like effects. The change in ARCI was assessed by the difference in measurements between baseline and 90 minutes after drink administration. Baseline was measure 15 minutes prior to capsule administration.
Time Frame: Measured 15 minutes prior to capsule administration and 90 minutes after drink administration
Population: Participants who completed all sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMP Arm | ALC Arm | THC Arm | AMP Placebo Arm | ALC Placebo Arm | THC Placebo Arm
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  ARC A | 2.96 (2.49) | 0.29 (2.44) | 0 (1.22) | -0.33 (0.76) | -0.58 (1.28) | -0.08 (1.02)
  ARC MBG | 3.67 (4.86) | -0.38 (2.45) | -0.83 (2.55) | -0.29 (0.86) | -1.29 (2.93) | -0.13 (0.95)
  ARC LSD | 1.08 (1.89) | 1.79 (1.93) | 1.42 (2.69) | -0.04 (0.95) | 0.29 (1.12) | 0.08 (0.93)
  ARC BG | 2.17 (2.39) | -2.54 (2.40) | -1.71 (2.03) | -1.29 (1.63) | -1.13 (1.57) | -0.67 (1.46)
  ARC PCAG | -1.21 (2.17) | 6.21 (2.92) | 3.54 (3.68) | 2.67 (2.96) | 1.92 (3.22) | 1.58 (1.91)
  ARC M | 2.63 (2.46) | 2.25 (2.51) | 2.04 (2.63) | 0.42 (0.97) | 0.13 (0.80) | 0.29 (0.62)

11. Primary Outcome: Change in Specific Drug Effects (Addiction Research Center Inventory) at 120 Minutes After Drink Administration
Description: Specific drug effects will be measured using the Addiction Research Center Inventory (Martin et al. 1971). The ARCI measures effects specific to drug classes, including the effects of AMP-like drugs (A scale, 0 to 11), morphine and benzedrine like drugs (MBG scale, 0 to 14), lysergic acid-like drugs (LSD scale, 0 to 14), benzedrine-like drugs (BG scale, 0 to 13), pentobarbital-chlorpromazine and ALC-like drugs (PCAG scale, 0 to 15), and cannabis-like drugs (M scale, 0 to 12). We used this questionnaire as a manipulation check to ensure that the drugs produced their typical drug-specific effects in this study. For example, zero value of A sacle would be minimum report of amphetamine-like drug effects, and 11 would be maximum report of amphetamine-like effects.The change in ARCI was assessed by the difference in measurements between baseline and 120 minutes after drink administration. Baseline was measure 15 minutes prior to capsule administration.
Time Frame: Measured 15 minutes prior to capsule administration and 120 minutes after drink administration
Population: Participants who completed all sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMP Arm | ALC Arm | THC Arm | AMP Placebo Arm | ALC Placebo Arm | THC Placebo Arm
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  ARC A | 2.17 (2.06) | -0.33 (1.34) | -0.08 (1.21) | -0.17 (0.70) | -0.71 (1.37) | -0.04 (0.86)
  ARC MBG | 3.33 (4.35) | -1.13 (2.13) | -0.96 (2.60) | -0.125 (0.85) | -1.29 (2.97) | -0.08 (0.65)
  ARC LSD | 0.38 (1.93) | 0.79 (1.28) | 1 (2.83) | -0.13 (1.15) | 0.04 (1.16) | -0.08 (0.93)
  ARC BG | 1.67 (2.12) | -2.04 (1.73) | -1.54 (1.64) | -1 (1.35) | -0.83 (1.55) | -0.38 (1.58)
  ARC PCAG | -1.08 (2.02) | 5.46 (2.93) | 2.88 (3.49) | 1.71 (2.65) | 1.63 (2.76) | 1.08 (1.98)
  ARC M | 1.83 (2.46) | 1.08 (1.56) | 1.42 (2.04) | 0.25 (0.85) | -0.04 (0.86) | 0.17 (0.56)

12. Primary Outcome: Change in Specific Drug Effects (Addiction Research Center Inventory) at 150 Minutes After Drink Administration
Description: Specific drug effects will be measured using the Addiction Research Center Inventory (Martin et al. 1971). The ARCI measures effects specific to drug classes, including the effects of AMP-like drugs (A scale, 0 to 11), morphine and benzedrine like drugs (MBG scale, 0 to 14), lysergic acid-like drugs (LSD scale, 0 to 14), benzedrine-like drugs (BG scale, 0 to 13), pentobarbital-chlorpromazine and ALC-like drugs (PCAG scale, 0 to 15), and cannabis-like drugs (M scale, 0 to 12). We used this questionnaire as a manipulation check to ensure that the drugs produced their typical drug-specific effects in this study. For example, zero value of A sacle would be minimum report of amphetamine-like drug effects, and 11 would be maximum report of amphetamine-like effects.The change in ARCI was assessed by the difference in measurements between baseline and 150 minutes after drink administration. Baseline was measure 15 minutes prior to capsule administration.
Time Frame: Measured 15 minutes prior to capsule administration and 150 minutes after drink administration
Population: Participants who completed all sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMP Arm | ALC Arm | THC Arm | AMP Placebo Arm | ALC Placebo Arm | THC Placebo Arm
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  ARC A | 2.29 (2.61) | -0.54 (1.14) | -0.17 (1.63) | -0.13 (0.69) | -0.54 (1.47) | -0.08 (0.83)
  ARC MBG | 2.96 (4.39) | -1.54 (1.96) | -0.96 (2.39) | 0.13 (0.76) | -1.25 (2.88) | -0.08 (0.88)
  ARC LSD | 0.5 (1.59) | 0.79 (1.35) | 0.58 (2.22) | 0.09 (1.08) | -0.13 (1.03) | -0.17 (0.82)
  ARC BG | 1.75 (2.31) | -2.04 (1.65) | -1.29 (1.86) | -0.43 (1.31) | -0.67 (1.24) | -0.42 (1.28)
  ARC PCAG | -1 (1.64) | 5.46 (2.95) | 2.58 (3.16) | 0.65 (2.17) | 1.58 (2.96) | 0.79 (1.79)
  ARC M | 1.54 (1.91) | 0.75 (1.33) | 0.83 (1.83) | 0.22 (0.74) | -0.21 (0.78) | 0.08 (0.41)

13. Primary Outcome: Change in Specific Drug Effects (Addiction Research Center Inventory) at 180 Minutes After Drink Administration
Description: Specific drug effects will be measured using the Addiction Research Center Inventory (Martin et al. 1971). The ARCI measures effects specific to drug classes, including the effects of AMP-like drugs (A scale, 0 to 11), morphine and benzedrine like drugs (MBG scale, 0 to 14), lysergic acid-like drugs (LSD scale, 0 to 14), benzedrine-like drugs (BG scale, 0 to 13), pentobarbital-chlorpromazine and ALC-like drugs (PCAG scale, 0 to 15), and cannabis-like drugs (M scale, 0 to 12). We used this questionnaire as a manipulation check to ensure that the drugs produced their typical drug-specific effects in this study. For example, zero value of A sacle would be minimum report of amphetamine-like drug effects, and 11 would be maximum report of amphetamine-like effects.The change in ARCI was assessed by the difference in measurements between baseline and 180 minutes after drink administration. Baseline was measure 15 minutes prior to capsule administration.
Time Frame: Measured 15 minutes prior to capsule administration and 180 minutes after drink administration
Population: Participants who completed all sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMP Arm | ALC Arm | THC Arm | AMP Placebo Arm | ALC Placebo Arm | THC Placebo Arm
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  ARC A | 1.58 (2.26) | -0.75 (1.19) | -0.21 (1.44) | -0.04 (0.91) | -0.33 (1.69) | -0.17 (1.13)
  ARC MBG | 1.92 (4.03) | -1.29 (1.88) | -0.67 (2.37) | 0.33 (1.24) | -1.08 (3.01) | -0.17 (0.82)
  ARC LSD | 0.46 (1.91) | 0.54 (1.02) | 0.54 (1.82) | 0.04 (1.04) | -0.04 (0.81) | 0.04 (0.95)
  ARC BG | 1.13 (2.15) | -1.5 (1.47) | -1.29 (1.78) | -0.33 (1.13) | -0.38 (1.41) | -0.29 (1.20)
  ARC PCAG | -0.46 (1.93) | 3.63 (3.01) | 2.13 (3.43) | 0.21 (2.50) | 0.71 (2.73) | 0.42 (1.59)
  ARC M | 1.21 (1.59) | 0.08 (1.02) | 0.71 (1.94) | 0.13 (0.68) | -0.13 (0.74) | -0.08 (0.28)

14. Primary Outcome: Change in Specific Drug Effects (Addiction Research Center Inventory) at 210 Minutes After Drink Administration
Description: Specific drug effects will be measured using the Addiction Research Center Inventory (Martin et al. 1971). The ARCI measures effects specific to drug classes, including the effects of AMP-like drugs (A scale, 0 to 11), morphine and benzedrine like drugs (MBG scale, 0 to 14), lysergic acid-like drugs (LSD scale, 0 to 14), benzedrine-like drugs (BG scale, 0 to 13), pentobarbital-chlorpromazine and ALC-like drugs (PCAG scale, 0 to 15), and cannabis-like drugs (M scale, 0 to 12). We used this questionnaire as a manipulation check to ensure that the drugs produced their typical drug-specific effects in this study. For example, zero value of A sacle would be minimum report of amphetamine-like drug effects, and 11 would be maximum report of amphetamine-like effects.The change in ARCI was assessed by the difference in measurements between baseline and 210 minutes after drink administration. Baseline was measure 15 minutes prior to capsule administration.
Time Frame: Measured 15 minutes prior to capsule administration and 210 minutes after drink administration
Population: Participants who completed all sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AMP Arm | ALC Arm | THC Arm | AMP Placebo Arm | ALC Placebo Arm | THC Placebo Arm
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
units on a scale
  ARC A | 1.0 (1.93) | -0.71 (1.20) | -0.46 (1.06) | -0.17 (0.82) | -0.54 (1.50) | 0.08 (1.21)
  ARC MBG | 1.38 (3.31) | -1.17 (2.08) | -0.88 (1.92) | 0.13 (1.15) | -0.79 (2.95) | 0.04 (0.86)
  ARC LSD | 0.63 (1.79) | 0.33 (0.92) | 0.54 (1.22) | 0.25 (0.90) | 1.67 (0.87) | 0.04 (1.04)
  ARC BG | 0.83 (1.61) | -1.25 (1.39) | -0.83 (1.40) | -0.17 (0.82) | -0.38 (1.06) | -0.13 (1.48)
  ARC PCAG | -0.29 (2.10) | 3.17 (3.17) | 1.04 (1.76) | -0.29 (1.43) | 0.21 (2.55) | 0.13 (1.68)
  ARC M | 0.96 (1.97) | 0.08 (0.97) | 0.21 (0.72) | 0 (0.42) | -0.17 (0.70) | -0.08 (0.28)

ADVERSE EVENTS:
Time Frame: During study only (1 Day)
Arm/Group | Healthy Adult Volunteers
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Adult Volunteers (N=28)
vomiting from alcohol dose (Gastrointestinal disorders) | 1 (1) — expected possible side effect of alcohol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No